CLINICAL TRIAL: NCT03577080
Title: The Effect of Adding Neuromuscular Electrical Stimulation to Endurance and Resistance Training on Exercise Capacity and Balance in Patients With Chronic Obstructive Pulmonary Disease: a Randomized Clinical Trial
Brief Title: Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Acheche Amal, principal investigator, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPD
Record Dates: First submitted 2018-06-05; First posted 2018-07-05 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: COPD
Keywords: COPD, Exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Differents groups received differents training protocoles during the same duration
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET+RT+ NMES (Active Comparator): neuromuscular electrical training NMES
  Interventions: Other: ET+RT+ NMES
- ET+RT (Placebo Comparator): placebo neuromuscular electrical training NMES
  Interventions: Other: ET+RT+ NMES

INTERVENTIONS:
Other: ET+RT+ NMES — Endurance training, resistance training and neuromuscular electrical stimuation were prformed. Intensity was gradually increased.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a preventable respiratory characterized by airflow obstruction that is not fully reversible. This disease a major cause of mortality worldwide. It is projected to rank the third-leading cause of death in 2020.

The objective of this study is to examine the effects of a physical therapy intervention in stable patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) patients have demonstrated important balance impairment (1).The deficit in balance control is identified as one of the risk factors of fall in subjects with COPD and alters their activities daily life (2,3). Porto and al. (2015) reported in a recent review that individuals with COPD have a decline in balance control when compared with healthy age matched controls(4).

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed by pulmonary function testing
* Clinically stable
* Abscence of other obstructive diseases
* Signed written consent
* Fall in the past five years or recent near fall

Exclusion Criteria:

* Neuromuscular diseases
* Severe psychiatric, neurologic or musculoskeletal conditions and /or instable cardiovascular diseases.
* Contre-indications to physical therapy
* Acute exacerbations a month before the intervention

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Balance outcomes | baseline
  The tests were performed using a stabilometric platform

SECONDARY OUTCOMES:
Pulmonary function test | baseline
  The test was performed using a Spirometry Zan 100 (Inspire Health GmbH, Germany)
Exercise tolerance | baseline
  The 6 minutes walk test
Force assesment | Baselline
  Maximal voluntary contraction (MVC) of the quadriceps muscle
Time Up and Go (TUG) | Baseline
  The patient initially sitting on an armless chair stand up walks 3 meters and returns and sit down again. The time was recorded
Berg Balance Scale (BBS) | Baseline
  The BBS contains 14 items. The score obtained from 0 to 56. from 0 to 20: high risk of falling , Above 56: No risk of falling

CONTACTS AND LOCATIONS:
Overall Officials: Amal Acheche, phd, Principal Investigator — Faculty of medecine Sousse
Locations (1):
- Research Unit of Exercise Physiology and Pathophysiology: from integral to molecular Biology, Medicine and Health (UR12 ES06) Faculty of Medicine of Sousse, Sousse, Tunisia

REFERENCES:
- [Result] Smith MD, Chang AT, Seale HE, Walsh JR, Hodges PW. Balance is impaired in people with chronic obstructive pulmonary disease. Gait Posture. 2010 Apr;31(4):456-60. doi: 10.1016/j.gaitpost.2010.01.022. Epub 2010 Mar 4. PMID 20206529
- [Result] Beauchamp MK, Hill K, Goldstein RS, Janaudis-Ferreira T, Brooks D. Impairments in balance discriminate fallers from non-fallers in COPD. Respir Med. 2009 Dec;103(12):1885-91. doi: 10.1016/j.rmed.2009.06.008. Epub 2009 Jul 9. PMID 19592229
- [Result] Roig M, Eng JJ, MacIntyre DL, Road JD, FitzGerald JM, Burns J, Reid WD. Falls in people with chronic obstructive pulmonary disease: an observational cohort study. Respir Med. 2011 Mar;105(3):461-9. doi: 10.1016/j.rmed.2010.08.015. PMID 20869227
- [Result] Porto EF, Castro AA, Schmidt VG, Rabelo HM, Kumpel C, Nascimento OA, Jardim JR. Postural control in chronic obstructive pulmonary disease: a systematic review. Int J Chron Obstruct Pulmon Dis. 2015 Jun 29;10:1233-9. doi: 10.2147/COPD.S63955. eCollection 2015. PMID 26170652